CLINICAL TRIAL: NCT04806022
Title: Effects of Different Forms of Fatigue on Double-Task Performance in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 21-PP-02
Record Dates: First submitted 2021-03-10; First posted 2021-03-19 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Fatigue Task first (Experimental): * First appointment :
    1. Pre-fatigue assessment
    2. mental fatigue task
    3. post-fatigue assessment
  * 7 resting days
  * second appointment
    1. Pre-fatigue assessment
    2. Muscle fatigue task
    3. post-fatigue assessment
  Interventions: Other: Fatigability assessment
- Muscle fatigue task first (Experimental): * First appointment :
    1. Pre-fatigue assessment
    2. Muscle fatigue task
    3. post-fatigue assessment
  * 7 resting days
  * second appointment
    1. Pre-fatigue assessment
    2. mental fatigue task
    3. post-fatigue assessment
  Interventions: Other: Fatigability assessment

INTERVENTIONS:
Other: Fatigability assessment — Each participant will do both types of fatigue over 2 appointments spaced by 7 days so that the subject can recover from induced fatigue. The sequence of fatigue tasks will be randomized.

SUMMARY:
The dual task (walking and cognitive task at the same time) is increasingly used in geriatrics in protocols for detecting people who are falling and/or for highlighting cognitive disorders. However, frail elderly people tend to get tired quickly and a lack of awareness of the effects of fatigue on dual-task performance could alter the diagnosis.

There are two types of fatigue: mental fatigue and peripheral muscle fatigue. Each participant will do both types of fatigue over 2 appointments spaced by 7 days so that the subject can recover from induced fatigue. The sequence of fatigue tasks will be randomized.

At the first appointment (day 0):

1. Pre-fatigue assessment :

   * The subject must walk on 10m with round trip for 1min.
   * the subject must do the arithmetic count of 3 in 3
   * Then comes the evaluation in double task (walking and counting at once for 1min). The subject must walk on 10m with round trip for 1min by doing the arithmetic count of 3 in 3 at the same time.
2. mental fatigue task or muscle fatigue task (randomized)
3. post-fatigue assessment (the same as pre-fatigue assessment)

7 resting days

Second appointment (day 7)

1. Pre-fatigue assessment :

   * The subject must walk on 10m with round trip for 1min.
   * the subject must do the arithmetic count of 3 in 3
   * Then comes the evaluation in double task (walking and counting at once for 1min). The subject must walk on 10m with round trip for 1min by doing the arithmetic count of 3 in 3 at the same time.
2. mental fatigue task or muscle fatigue task (randomized)
3. post-fatigue assessment (the same as pre-fatigue assessment)

ELIGIBILITY:
Young group

Inclusion Criteria:

* 20 to 40 years old

Exclusion Criteria:

* psychiatric disorders
* Severe hearing or vision loss
* Motor or sensory disability that may interfere with test completion

Old group

Inclusion Criteria:

* 65 to 90 years old
* less than 3 Fried's criteria of fragility
* walking ability without technical assistance (at least 10m).

Exclusion Criteria:

* psychiatric disorders
* Severe hearing or vision loss
* Motor or sensory disability that may interfere with test completion

Old frail group

Inclusion Criteria:

* 65 to 90 years old
* 3 or more Fried's criteria of fragility
* walking ability without technical assistance (at least 10m).

Exclusion Criteria:

* psychiatric disorders
* Severe hearing or vision loss
* Motor or sensory disability that may interfere with test completion

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Dual task performance after muscular fatigue | at inclusion (day 0)
  Dual task performance (DTEspeed motor performance; DTEcog cognitive performance) will be compared before and after a protocol of peripheral mental and muscular fatigue.
  For Dual Task Performance, the cognitive task performance (maximum count count - error count) performed alone (single ST task) and performed while walking (double ST task) will be compared.
Dual task performance after cognitive fatigue | at day 7
  Dual task performance (DTEspeed motor performance; DTEcog cognitive performance) will be compared before and after a protocol of peripheral mental and muscular fatigue.
  For Dual Task Performance, the cognitive task performance (maximum count count - error count) performed alone (single ST task) and performed while walking (double ST task) will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GUERIN, Principal Investigator — Nice University Hospital, Gerontology Department
Locations (1):
- CHU de Nice, Nice, France